CLINICAL TRIAL: NCT04500054
Title: The Effects Of Music Listening In Patients Undergoing Retrograde Intrarenal Surgery On Basic Life Findings, Anxiety, Pain, And The Amount Of Analgesic Used.
Brief Title: The Effects Of Music In Retrograde Intrarenal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeliz Ciğerci, Assistant Proffesor PhD, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: (2019/165
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Retrograde Intrarenal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention Group (Experimental): The music intervention group listened to the music by the researchers for the duration of 15 minutes one hour before the surgery as well as the standard care.
  Interventions: Other: Music Listening
- No Intervention Group (No Intervention): The control group patients received standard care only.

INTERVENTIONS:
Other: Music Listening — The music type was chosen by the patients and researchers did not have any influence on their choices.
  Arms: Music Intervention Group

SUMMARY:
This study aimed to investigate the effect of music listening during the preoperative and postoperative stages in patients undergoing retrograde intrarenal surgery(RIRS) on basic life findings, anxiety, pain, and the amount of analgesic used. This is a randomized controlled experimental study.

The study was conducted with two groups: the intervention group (n=30) and control group (n=30). The control group received standard care. In contrast, the intervention group, in addition to standard care, was listened to the music by the researchers for 15 minutes one hour before their surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above,
* had elective RIRS,
* without hearing/speech impairment,
* without mental problems,
* without a diagnosis of psychiatric disorders,
* without a diagnosis of depression,
* had the surgery under general anesthesia,
* and volunteered to participate.

Exclusion Criteria:

* Patients under 18 years of age,
* with hearing/speech impairment,
* with mental problems,
* with a diagnosis of psychiatric disorders,
* with a diagnosis of depression,
* undergoing the surgery through spinal anesthesia,
* not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Anxiety (VAS-A) | 2 days
  VAS-A is a 10 cm long measuring instrument with the score range from 0 to 10 with 0 points showing "no anxiety" and 10 points showing "I feel a lot of anxiety" .

SECONDARY OUTCOMES:
Visual Analog Scale for Pain (VAS) | 1 day
  VAS scale is a single-dimensional scale that is commonly used to evaluate pain severity. According to VAS, pain intensity is rated as "no pain" with 0 points, and "the most severe pain imaginable" with 10 points. Pain intensity ranges were determined by VAS as follows; mild pain below 3 points, as moderate pain between 3 and 6 points, and as severe pain above 6 points.The VAS pain scale was applied to the patients once on the first postoperative day, for the level of pain they felt.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No